CLINICAL TRIAL: NCT04833816
Title: Ketamine Low dOse Evaluation on Morphine Consumption in Traumatic Patient
Acronym: KLOE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-48; 2020-004812-81 (EudraCT Number)
Record Dates: First submitted 2021-04-05; First posted 2021-04-06 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Traumatic Injury
Keywords: ketamine; analgesia; ISS; trauma
MeSH Terms: conditions — Wounds and Injuries; Agnosia | interventions — Administration, Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamin (Experimental): Patient will get a bolus of ketamine at 0.1 mg / kg followed by a continuous infusion of ketamine at a dose of 0.15 mg / kg / hour
  Interventions: Drug: Administration of drug
- Placebo (Placebo Comparator): Patient will get a bolus of NaCL at 0.1 mg / kg followed by a continuous infusion of NaCl at a dose of 0.15 mg / kg / hour
  Interventions: Drug: Administration of drug

INTERVENTIONS:
Drug: Administration of drug — Administration of ketamin during the 48h after trauma

SUMMARY:
The aim of this study is to demonstrate a significant reduction of at least 25% in opioid consumption at 48 hours of management of severe trauma, while demonstrating non-inferiority in terms of analgesia, in a group of patients receiving a continuous infusion of low dose ketamine compared to a placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult
* Trauma patient presenting at least 2 lesions in two different regions as defined by the ISS (injury severity score) (Head or neck, Face, Thorax, Abdomen and pelvic contents, Upper limbs or pelvic girdle, Lower limbs, External (any skin surface).
* Patient presenting at least two regional disorders classified as moderate to maximum defined by an AIS (Abbreviated Injury Scale)> 1.
* Patient having signed an informed consent

Exclusion Criteria:

* Patients with an indication for deep sedation (intracranial hypertension or acute respiratory distress syndrome).
* Patient in whom the infusion could not be started within the first 6 hours of initial treatment.
* Patient whose state of consciousness is incompatible with understanding the protocol.
* Patient with chronic unbalanced arterial hypertension.
* Patient with severe heart failure.
* Patient with a BMI> 35 kg / m² or a weight of more than 120 kg.
* Patient with chronic analgesic consumption defined by consumption of opioid derivatives for more than a week for an intercurrent illness.
* Presence of a history of chronic pain.
* Presence of a history of epilepsy.
* Presence of a history of psychosis or drug addiction.
* Presence of a history of stroke.
* Patients with an allergy to the molecule or excipients composing ketamine
* Patients with an allergy to the molecule or to the excipients making up sufentanil or paracetamol.
* Pregnant or breastfeeding woman.
* Patient not understanding French.
* Protected adult patient (under guardianship, curatorship or legal protection).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2025-10-04 (Actual); Study Completion 2026-01-03 (Actual)

PRIMARY OUTCOMES:
Total dose of sufentanil | 48 hours
  All doses of sufentanil and opiods administration

SECONDARY OUTCOMES:
Total amount of opiods | 5 days
Pain assessment | 5 days
Delirium | 5 days
  Scale CAM-ICU (confusion assesment method)
Global Quality of life | 3 months
  SF-36 score
Chronical pain | 3 months
  SF-MPQ-2

CONTACTS AND LOCATIONS:
Overall Officials: Jean Olivier ARNAUD, Study Director — AP-HM
Locations (1):
- Service Anesthésie Réanimation - Hôpital nord, Marseille, France

IPD SHARING:
Plan to Share IPD: No